CLINICAL TRIAL: NCT01970683
Title: Effect of Perioperative Probiotics on Clinical Outcomes of Patients Undergoing Major Abdominal Operation in Community Settings.
Brief Title: Probiotics and Recovery From Surgery
Acronym: PROGRESS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: organizational problems
Sponsor: Catholic Health Initiatives (Other)
Responsible Party: Principal Investigator, Jan Franko, Surgical Oncologist, Catholic Health Initiatives
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: MMC-2013-132
Record Dates: First submitted 2013-10-23; First posted 2013-10-28 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Major Abdominal Operation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- VSL #3 (Experimental): probiotics given orally BID
  Interventions: Dietary Supplement: VSL #3 BID
- placebo (Other): Near-identically appearing placebo
  Interventions: Dietary Supplement: VSL #3 BID

INTERVENTIONS:
Dietary Supplement: VSL #3 BID

SUMMARY:
The study will investigate whether probiotics given just before and shortly after major abdominal operation improve outcomes.

DETAILED DESCRIPTION:
Perioperative probiotic intervention is associated with approximately 30% reduction of primary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* All elective major GI surgical patients

Exclusion Criteria:

* • Current episode of acute pancreatitis as defined by clinician

  * Active medication-induced immunosuppression including systemic corticosteroids, chemotherapy within 4 weeks, immunomodulating agents with transplant indication, biologicals for rheumatoid arthritis and inflammatory bowel disease. Topical chemotherapy or corticosteroids, and chemotherapy applied during operation are allowed.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2014-08; Primary Completion 2017-02 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
30-day postsurgical outcome including death, infection, readmission | within 30 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Mercy Medical Center-Des Moines, Des Moines, Iowa, United States

REFERENCES:
- [Derived] Franko J, Raman S, Krishnan N, Frankova D, Tee MC, Brahmbhatt R, Goldman CD, Weigel RJ. Randomized Trial of Perioperative Probiotics Among Patients Undergoing Major Abdominal Operation. J Am Coll Surg. 2019 Dec;229(6):533-540.e1. doi: 10.1016/j.jamcollsurg.2019.09.002. Epub 2019 Sep 25. PMID 31562911